CLINICAL TRIAL: NCT06259266
Title: Catheter Dysfunction Rate in Patients Undergoing Kidney Replacement Therapy. Evaluation of the Safety and Efficacy of Anti-reflux Valves Without Heparin Lock Solution
Acronym: DUKE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Abandonment of financial partners
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire HEMOTECH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0171; 2012-A00530-43
Record Dates: First submitted 2013-11-26; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2013-11

CONDITIONS: Chronic Renal Failure; Haemodialysis, Haemodiafiltration, Haemofiltration; Kidney Replacement Therapy; Catheter Infection, Catheter Dysfunction, Catheter Related Bloodstream Infections
Keywords: Catheter infection, catheter dysfunction, catheter related bloodstream infections,
MeSH Terms: conditions — Kidney Failure, Chronic

ARMS (2):
- valce arm (Experimental): Two strategies are compared in a parallel plan : a "valve arm " (implementation of TEGO ® valve associated with interdialytic saline locks) and a "control arm" ( standard care ).
  Interventions: Other: Anti-reflux valve for dialysis catheter
- control arm (Other): Two strategies are compared in a parallel plan : a "valve arm " (implementation of TEGO ® valve associated with interdialytic saline locks) and a "control arm" ( standard care ).
  Interventions: Other: Anti-reflux valve for dialysis catheter

INTERVENTIONS:
Other: Anti-reflux valve for dialysis catheter

SUMMARY:
Catheter dysfunction and infections are the most common complications observed among patients with dialysis catheters for long-term dialysis ( CDLD ) . They are causing a worsening of the morbidity and mortality of patients , loss of quality of renal replacement therapy , a reduction in the duration of catheterization , as well as increased spending related to health care.

The use of anti- reflux ( Tego ® , ICU Medical , USA, distributed by the Laboratory Hemotech , FRANCE ) valves reduces the rate of dysfunction and infections CDLD( catheters for long-term dialysis ). Unpublished preliminary data suggest that these valves allow parallel use of interdialytic saline locks without increasing the risk of dysfunction. This strategy would therefore achieve significant savings usual interdialytic CDLD( catheters for long-term dialysis )locks ( including heparin) whose use is not devoid of potentially serious adverse events and whose health care costs have increased dramatically in recent years . Moreover, this would also produce savings in fibrinolytic treatment.

A randomized controlled trial is needed to assess the effectiveness of TEGO ® valves in combination with saline locks on the risk of dysfunction CDLD(catheters for long-term dialysis ) .

DETAILED DESCRIPTION:
Interventional prospective, multicenter (8 dialysis units) , randomized, controlled, open study. Two strategies are compared in a parallel plan : a "valve arm " (implementation of TEGO ® valve associated with interdialytic saline locks) and a "control arm" ( standard care ). Rate of dialysis session with dysfunctions during the first six months of the study is the primary endpoint. It will be analyzed " per protocol ". The total duration of patient follow-up is 12 months.

After the first 6 months, patients in the "valve arm" retain the same type of care until the end of the study. The control patients continue to receive the usual concentrated heparin locks . The secondary endpoints of the study will be analyzed to 12 months. Training of health care teams is expected before the start of the study .

ELIGIBILITY:
Inclusion Criteria:

* Haemodialysis patients

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Rate of dialysis session with dysfunctions | during the first six months

SECONDARY OUTCOMES:
evaluation of the infectious complications associated with CDLD (catheters for long-term dialysis) | during the first six months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Elisabeth HENG, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de CERMONT-Ferrand, Clermont-Ferrand, France